CLINICAL TRIAL: NCT07243587
Title: Cohort of the Franco-European Multidisciplinary Institute of Endometriosis
Acronym: IFEMEndo
Status: Recruiting | Type: Observational
Sponsor: Clinique Tivoli Ducos (Other)
Responsible Party: Sponsor
Other Study IDs: Cli-Tiv-01-2021
Record Dates: First submitted 2021-06-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Endometriosis; Deep Endometriosis; Pelvic Pain
Keywords: cohort; prospective
MeSH Terms: conditions — Endometriosis; Pelvic Pain | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: OBSERVATIONAL — OBSERVATIONAL STUDY

SUMMARY:
Endometriosis is a chronic benign gynecological condition affecting 5 to 10% of women of reproductive age, often responsible for pelvic pain, digestive symptoms, and infertility, leading to a significant reduction in quality of life. Despite its high prevalence, the long-term outcomes of different medical and surgical treatments remain poorly documented.

The IFEMENDO study is a prospective, observational, single-center, non-interventional cohort conducted at the Endometriosis Center of Clinique Tivoli-Ducos in Bordeaux, France. The objective is to evaluate the long-term efficacy of various therapeutic strategies-both medical and surgical-in terms of symptom improvement, quality of life, recurrence, and fertility outcomes.

Women with histologically or radiologically confirmed pelvic endometriosis are invited to participate. Data are collected through standardized questionnaires at baseline and at 1, 3, 5, 7, and 10 years after inclusion, either via the secure NO ENDO online platform or in paper form. The study will contribute to a better understanding of the natural history of endometriosis and the long-term effectiveness of different treatment approaches, ultimately supporting improvements in clinical management and patient care.

DETAILED DESCRIPTION:
Detailed Description

The IFEMENDO study is an observational, single-center, non-interventional, prospective cohort conducted at the Endometriosis Center of Clinique Tivoli-Ducos in Bordeaux, France. The study aims to evaluate the long-term efficacy of various medical and surgical treatments for deep pelvic endometriosis in terms of symptom improvement, quality of life, recurrence rate, and fertility outcomes.

Endometriosis is a benign but chronic gynecological condition affecting 5 to 10% of women of reproductive age, most of whom are professionally active. It can cause pelvic pain of varying duration and intensity, digestive dysfunction, and infertility, leading to significant deterioration in quality of life and social well-being. Diagnosis is often delayed for several years after symptom onset, which explains the high prevalence of advanced stages and deep localizations at the time of diagnosis. Despite its frequency, the natural history of endometriosis and long-term outcomes after treatment remain poorly documented. Existing studies are mostly randomized trials with small sample sizes or retrospective series from single surgical teams, with follow-up rarely exceeding two or three years.

This study will include all women with histologically or radiologically confirmed pelvic endometriosis seen in consultation or operated on at the Endometriosis Center. After obtaining non-opposition consent, each participant will complete a baseline questionnaire including medical and surgical history, endometriosis-related symptoms, fertility status, and quality of life. In the case of surgery, the surgeon will complete a detailed form describing disease localization, surgical procedures performed, and any postoperative complications.

Participants will then be invited to complete follow-up questionnaires at 1, 3, 5, 7, and 10 years after inclusion. These follow-up questionnaires will cover the same domains: symptoms, fertility, and quality of life. Data will be collected through the secure NO ENDO online platform or, if preferred, on paper forms later transcribed into the electronic database by trained clinical research associates.

Registry Procedures and Quality Assurance

A quality assurance plan has been implemented to ensure the validity, reliability, and completeness of data collected in the registry. Data validation procedures include automated range and consistency checks at the time of data entry, as well as periodic manual reviews. Source data verification will be performed by comparing data entered in the NO ENDO system against medical records and operative reports.

Standard Operating Procedures are in place to guide all registry activities, including patient recruitment, informed consent documentation, data entry and management, monitoring, adverse event reporting, and database updates. The registry complies with French data protection regulations and the European General Data Protection Regulation.

Sample Size and Data Management

All eligible women consulting at the Endometriosis Center and meeting inclusion criteria will be invited to participate. The expected cohort size is several thousand patients, allowing robust statistical analyses over a 10-year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Women aged >18 years
* Women with histologically or radiologically confirmed deep endometriosis (and/or) infiltrating the colon and/or rectum
* Women affiliated with the social security system

Exclusion Criteria:

* Refusal to participate
* Patients under guardianship or curatorship, or deprived of liberty

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with deep endometriosis infiltrating the colon and / or the rectum
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2036-02 (Estimated); Study Completion 2036-02 (Estimated)

PRIMARY OUTCOMES:
Efficacity of differents treatments | Each patient fills out the questionnaires at inclusion, and then at 1 year, 3 years, 5 years, 7 years, and 10 years.
  The primary objective is to study the long-term efficacy of different treatments, both drug and surgical, in terms of symptom improvement: change in patient-reported symptom scores over time (unit: score on a validated symptom scale).
Efficacity of differents treatments | Each patient fills out the questionnaires at inclusion, and then at 1 year, 3 years, 5 years, 7 years, and 10 years.
  The primary objective is to study the long-term efficacy of different treatments, both drug and surgical, in terms of quality of life: changes in quality of life scores over time (unit: points on a validated QoL questionnaire).
Efficacity of differents treatments | Each patient fills out the questionnaires at inclusion, and then at 1 year, 3 years, 5 years, 7 years, and 10 years.
  The primary objective is to study the long-term efficacy of different treatments, both drug and surgical, in terms of recurrence rate: proportion of patients experiencing recurrence of the condition during follow-up (unit: percentage).
Efficacity of differents treatments | Each patient fills out the questionnaires at inclusion, and then at 1 year, 3 years, 5 years, 7 years, and 10 years.
  The primary objective is to study the long-term efficacy of different treatments, both drug and surgical, in terms of taux de grossesse : the proportion of patients who achieved a pregnancy during follow-up (unit: percentage).

SECONDARY OUTCOMES:
Evaluation of digestive function | Each patient fills out the questionnaires at inclusion, and then at 1 year, 3 years, 5 years, 7 years, and 10 years.
  To evaluate digestive function, before and after treatment of digestive endometriosis compared to different colorectal surgery techniques in deep endometriosis
Evaluation of the probability of pregnancy | Each patient fills out the questionnaires at inclusion, and then at 1 year, 3 years, 5 years, 7 years, and 10 years.
  To evaluate the probability of pregnancy after different techniques of management of endometriosis of the ovaries, in order to assess their impact on ovarian reserve and the chances of pregnancy after treatment
Evaluation of the risk factor | Each patient fills out the questionnaires at inclusion, and then at 1 year, 3 years, 5 years, 7 years, and 10 years.
  To study the risk factors present in the patients' history and having a relationship with the appearance of different specific localizations of the disease
Evaluation of evolution of endometriosis | Each patient fills out the questionnaires at inclusion, and then at 1 year, 3 years, 5 years, 7 years, and 10 years.
  To study prospectively the evolution of endometriosis, with or without treatment, and the predictive factors for the development of severe forms and deep localizations of pelvic endometriosis

CONTACTS AND LOCATIONS:
Locations (1):
- Clinique Tivoli Ducos, Bordeaux, France

IPD SHARING:
Plan to Share IPD: Undecided